CLINICAL TRIAL: NCT03076424
Title: Is Weight Change and Glucoregulation Related to Dietary Intake, the Gut Microbiome or the Interaction Between The Two Variables?
Brief Title: The Effect of Nutrient Intake on the Microbiome, Weight, and Glucoregulation (NI-MWG)
Acronym: NI-MWG
Status: Completed | Type: Observational
Sponsor: North Dakota State University (Other)
Collaborators: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, Pharm. D., Ph.D., North Dakota State University
Other Study IDs: NDSU-PS
Record Dates: First submitted 2017-02-22; First posted 2017-03-10 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Type2 Diabetes
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma/serum samples and fecal samples will be collected from each patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Obese patients (BMI greater than or equal to 30 kg/m2) with Type 2 Diabetes Mellitus.
  Interventions: Other: no intervention used
- 2: Obese patients (BMI greater than or equal to 30 kg/m2) without Type 2 Diabetes Mellitus.
  Interventions: Other: no intervention used
- 3: Normal weight lean controls without Type 2 Diabetes Mellitus.
  Interventions: Other: no intervention used

INTERVENTIONS:
Other: no intervention used — Patients will be giving a blood sample after 8 hours of fasting.

SUMMARY:
The purpose of this study is to investigate a persons dietary intake and its effect on the gut microbiome and the association of those two variables on weight and glucoregulation. Specifically, the investigators will compare the gut microbiota, fasting glucose and insulin, c-peptide and hemoglobin A1-c in three groups of subjects: obese patients (BMI ≥ 30 kg/m2) with type 2 diabetes mellitus (T2DM), obese patients without T2DM, and normal weight lean controls without T2DM. Each patient will also complete a detailed dietary recall (ASA-24) to investigate the association with diet, microbiome and weight/glucoregulation.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18-65 (inclusive, at time of informed consent)
3. BMI ≥ 30 kg/m2 with T2DM
4. BMI ≥ 30 kg/m2 without T2DM
5. Normal weight lean controls without T2DM

Exclusion Criteria:

1. Tobacco use in past three months - will add unnecessary confound to the data.
2. Taking a medication on a routine/recent basis which is known to significantly influence gastrointestinal transit time or affect the microbiome or other variables significantly (as determined by study pharmacist/MD)
3. Has taken an oral or injectable antibiotic in the past 3 months
4. Has taken a commercially prepared probiotic and/or prebiotic agent in the 3 months
5. History of significant intestinal disease or disorder (e.g., crohn's disease, ulcerative colitis)
6. History of gastrointestinal surgery that may impact measures of biological variables, as determined by the investigator
7. Medical condition expected to impact the biological variables of interest or interfere with providing a sample, as determined by the investigator.
8. Unable to speak/read English
9. Breastfeeding, pregnant, or planning to become pregnant within the duration of the study as assessed through self-report on medical history
10. Unwilling to use a medically acceptable form of contraception during study involvement. Medically acceptable forms of contraception include oral contraception, physical barrier methods and/or abstinence.
11. Any known infectious disease such as Viral Hepatitis or HIV (as determined by study pharmacist/MD)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese diabetics, obese non-diabetics and controls
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Intestinal Microbiome Composition | One sample collected upon study enrollment
  The ratio of firmicutes to bacteroidetes will be the primary focus of the microbiome evaluation.

SECONDARY OUTCOMES:
Fasting Glucose | One sample collected upon study enrollment
  Serum glucose (fasting) will be measured from collected blood sample and compared between the 3 subject groups.
Fasting Insulin | One sample collected upon study enrollment
  Plasma insulin (fasting) will be measured from collected blood sample and compared between the 3 subject groups.
C-peptide | One sample collected upon study enrollment
  c-peptide will be measured from collected blood sample and compared between the 3 subject groups.
Hemoglobin A1-c | One sample collected upon study enrollment
  hemoglobin A1-c will be measured from collected blood sample and compared between the 3 subject groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuropsychiatric Research Institute (NRI), Fargo, North Dakota, United States